CLINICAL TRIAL: NCT01499979
Title: In Situ Hypothermic Perfusion During Right Hemihepatectomy
Brief Title: Hypothermic Perfusion During Hemihepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Megan J. Reiniers, PhD student, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011_214; NL37241.018.11 (Other: Centrale Commissie Mensgebonden Onderzoek (CCMO))
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Ischemia-reperfusion Injury
Keywords: Ischemia-reperfusion injury; In situ hypothermic perfusion; In situ hypothermic preservation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vascular inflow occlusion (No Intervention): Patients that will receive intermittent vascular inflow occlusion, the standard method for vascular occlusion at our institution, during liver resection.
- Hypothermic perfusion (Experimental): Patients will receive in situ hypothermic perfusion of the future remnant liver during liver resection.
  Interventions: Procedure: In situ hypothermic perfusion

INTERVENTIONS:
Procedure: In situ hypothermic perfusion — In situ perfusion of the future remnant liver with chilled lactated Ringer's solution during liver resection.
  Other Names: In situ hypothermic preservation
  Arms: Hypothermic perfusion

SUMMARY:
Rationale

Currently, hepatic resection is often the only curative treatment for primary or secondary hepatic malignancies and is also frequently performed in patients with benign liver tumors to prevent malignant transformation and/or alleviate symptoms. Liver resections are nowadays associated with low mortality and acceptable morbidity. As result of that, an increasing number of patients is currently under consideration for resection of more complex or large tumors, thus requiring extensive resection procedures. Application of vascular exclusion (i.e., clamping of the portal vein and hepatic artery) during such procedures reduces blood loss, which is one of the most important factors affecting peri-operative outcomes. However, vascular exclusion leads to ischemia-reperfusion (I/R) injury as an inevitable side-effect, which adversely impacts postoperative liver function and regeneration. Additional cooling of the liver by means of hypothermic perfusion is expected to further reduce intraoperative blood loss, as well as to protect the liver from I/R injury. Therefore, the aim of this pilot study is to cool the future remnant liver (FRL) in situ during right hemihepatectomy under vascular exclusion. Consequently, an overall improvement in postoperative outcomes is expected due to a decrease in intraoperative blood loss, reduced parenchymal damage, and a better ability of the liver remnant to regenerate.

Objective

To reduce intraoperative blood loss and enhance tolerance of the FRL to I/R injury during right hemihepatectomy under vascular exclusion by means of in situ hypothermic perfusion with retrograde outflow (R-IHP) of the FRL.

Study design

The study is designed as a prospective randomized pilot study in 18 patients (9 interventions and 9 controls) to assess the effects of the proposed intervention. Additionally, 4 patients will be included separately for assessment of the intervention's feasibility prior to randomized inclusion.

Study population

Eligible patients for participation in this study are those planned to undergo right hemihepatectomy under vascular inflow occlusion because of a malignant or benign liver tumor, and who do not suffer from any hepatic co-morbidity that might influence postoperative outcomes (i.e., severe steatosis, cholestasis, cirrhosis, or hepatitis B/C infection).

Intervention

During right hemihepatectomy, the FRL of patients allocated to the intervention group will be perfused with a chilled perfusion solution (i.e., lactated Ringer's solution).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for right hemihepatectomy under vascular inflow occlusion for a malignant or benign hepatic tumor
* Diagnostic exclusion of hepatic co-morbidity, that is:

  * Cirrhosis,
  * Severe steatosis (≥ 30%),
  * Cholestasis, and
  * Hepatitis B/C infection
* Age ≥ 18 years
* Signed informed consent obtained prior to any study-specific procedure
* ASA classification I-III

Exclusion Criteria:

* Patients diagnosed with any of the hepatic co-morbidities listed under point 2 of the inclusion criteria
* Age < 18 years
* BMI > 35 kg/m2
* ASA classification IV/V
* Patient is scheduled for a combined surgical procedure (e.g., bile duct resection, gastrointestinal procedures)
* Patient underwent liver resection ≤ 1 year prior to scheduled surgery
* Emergency operations
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Postoperative hepatocellular damage | 5 days postoperatively
  Hepatocellular damage expressed as an postoperative increase in transaminases (i.e., AST and ALT).

SECONDARY OUTCOMES:
Intraoperative blood loss | 2-3 hours
  Blood loss during surgery
Postoperative complications | 5 days postoperatively
  Incidence of surgery-related complications
Regeneration of liver function and volume | 3 days
  Regeneration of liver function (measured via hepatobiliary scintigraphy) and -volume (measured via CT volumetry).

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Thomas M. van Gulik, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Megan J. Reiniers, MSc, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Rowan F. van Golen, MSc, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center (AMC), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azoulay D, Eshkenazy R, Andreani P, Castaing D, Adam R, Ichai P, Naili S, Vinet E, Saliba F, Lemoine A, Gillon MC, Bismuth H. In situ hypothermic perfusion of the liver versus standard total vascular exclusion for complex liver resection. Ann Surg. 2005 Feb;241(2):277-85. doi: 10.1097/01.sla.0000152017.62778.2f. PMID 15650638
- [Background] Dinant S, van Veen SQ, Roseboom HJ, van Vliet AK, van Gulik TM. Liver protection by hypothermic perfusion at different temperatures during total vascular exclusion. Liver Int. 2006 May;26(4):486-93. doi: 10.1111/j.1478-3231.2006.01248.x. PMID 16629653
- [Background] Verhoef C, de Wilt JH, Brunstein F, Marinelli AW, van Etten B, Vermaas M, Guetens G, de Boeck G, de Bruijn EA, Eggermont AM. Isolated hypoxic hepatic perfusion with retrograde outflow in patients with irresectable liver metastases; a new simplified technique in isolated hepatic perfusion. Ann Surg Oncol. 2008 May;15(5):1367-74. doi: 10.1245/s10434-007-9714-z. Epub 2008 Feb 1. PMID 18239976
- [Result] Reiniers MJ, van Golen RF, Heger M, Mearadji B, Bennink RJ, Verheij J, van Gulik TM. In situ hypothermic perfusion with retrograde outflow during right hemihepatectomy: first experiences with a new technique. J Am Coll Surg. 2014 Jan;218(1):e7-16. doi: 10.1016/j.jamcollsurg.2013.09.013. Epub 2013 Nov 6. No abstract available. PMID 24210146